CLINICAL TRIAL: NCT02305186
Title: A Randomized Multicenter Ib/II Study to Assess the Safety & Immunological Effect of Chemoradiation Therapy in Combination With Pembrolizumab Compared to CRT Alone Resectable/Borderline Resectable Pancreatic Cancer
Brief Title: Safety and Immunological Effect of Pembrolizumab in Resectable or Borderline Resectable Pancreatic Cancer
Acronym: UVA-PC-PD101
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Craig L Slingluff, Jr (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Director of the UVA Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17801
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
Keywords: Immunotherapy; Neoadjuvant; Resectable; Borderline resectable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neodjuvant CRT + Pembrolizumab (Experimental): Standard neoadjuvant chemoradiation treatment (CRT) with pembrolizumab
  Interventions: Drug: Pembrolizumab; Radiation: Neoadjuvant Chemoradiation
- Neoadjuvant CRT (Active Comparator): Standard neoadjuvant chemoradiation treatment (CRT) alone
  Interventions: Radiation: Neoadjuvant Chemoradiation

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered at a dose of 200 mg IV every 3 weeks on days 1, 22, and 43 during concurrent neoadjuvant chemoradiation treatment
  Other Names: MK-3475; Keytruda
  Arms: Neodjuvant CRT + Pembrolizumab
Radiation: Neoadjuvant Chemoradiation — Chemoradiation with capecitabine (825 mg/m2 orally twice daily, Monday through Friday, on days of radiation only) and radiation (50.4 Gy in 28 fractions over 28 days)

SUMMARY:
The purpose of this clinical trial is to study an experimental drug called pembrolizumab or MK-3475 for use in combination with chemotherapy and radiation therapy for patients with resectable (surgical removal) or borderline resectable pancreatic cancer. In general, pancreatic cancer that cannot be removed by surgery is sometimes treated with chemotherapy and radiation therapy, called neoadjuvant treatment, to shrink the tumor so that surgery might be possible. However, this is not always effective at shrinking the tumor enough to allow it to be removed with surgery. Recent discoveries suggest that the investigators own immune system might have a role in controlling the growth of tumors. Drugs such as pembrolizumab can stimulate the immune system against cancer. The purpose of this study is to investigate whether pembrolizumab can be used safely during neoadjuvant treatment and can improve the body's immune response against pancreatic cancer.

Pembrolizumab has been approved for treatment of patients with melanoma but has not been proven to be safe or helpful in patients with pancreatic cancer and is not approved by the U.S. Food and Drug Administration (FDA) for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.
2. Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
3. Adequate organ function
4. In subjects requiring biliary decompression, metal stent or drainage using percutaneous transhepatic cholangiogram (PTC) are allowed

Exclusion Criteria:

1. Immunodeficiency or taking steroid or any other form of immunosuppressive therapy
2. Has a plastic biliary stent for decompression
3. Metastatic disease
4. Prior treatment for pancreatic cancer (other than 4-8 cycles of Folfirinox) or prior treatment with radiation for other diagnoses to the expected pancreatic cancer treatment area
5. Active autoimmune disease
6. Pregnancy or Nursing
7. Known history of Human Immunodeficiency Virus (HIV) or Hepatitis B or C
8. Prior monoclonal antibody within 4 weeks prior to study Day 1
9. Known additional malignancy that is progressing or requires active treatment
10. Evidence of interstitial lung disease or active, non-infectious pneumonitis
11. Active infection requiring systemic therapy
12. Prior therapy with an anti-Program Death (PD-1) antibody, anti-PD-L1, anti-PD-L2, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of Tumor Infiltrating Lymphocytes (TILs) per high powered field (hpf) in pancreatic tissue (resected tissue). | 2-3 years
Safety: Incidence of Dose-Limiting Toxicities (DLTs) | 2-3 years

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 2-4 years
Overall survival (OS) | 2-4 years
Response Rate (RR) | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Osama Rahma, MD, Study Chair — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Hartford HealthCare, Hartford, Connecticut
  - University of Miami, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia